CLINICAL TRIAL: NCT02154607
Title: Clinical Trial Analyzing the Impact of Continuous Defocused CO2 Laser Vaporisation on the Histological Malignant Transformation of Erosive Oral Lichen Planus
Brief Title: Impact of Continuous Defocused CO2 Laser Vaporisation on the Histological Malignant Transformation of Erosive Oral Lichen Planus in Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TechnischeUM
Record Dates: First submitted 2014-03-27; First posted 2014-06-03 (Estimated); Last update posted 2014-06-03 (Estimated); Status verified 2014-05

CONDITIONS: Oral Lichen Planus
Keywords: oral lichen planus; recurrence; Treatment; cancer; Primary disease Management
MeSH Terms: conditions — Lichen Planus, Oral; Recurrence; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Symptomatic treatment (No Intervention): Symptomatic analgetic Treatment only was performed without any Manipulation of OLP lesions.
- CO2-Laser Treatment (Active Comparator): CO2-Laser Vaporisation was performed of OLP lesions under local anaesthesia.
  Interventions: Device: CO2-Laser Treatment

INTERVENTIONS:
Device: CO2-Laser Treatment
  Arms: CO2-Laser Treatment

SUMMARY:
Oral Lichen Planus (OLP) is a common condition with its erosive variant occasionally presenting a management challenge to the clinician. In addition it can have debilitating consequences on the patients' quality of life. The malignant transformation of OLP has been well documented. The aims of this work were to measure the number of patients developing malignant transformationof OLP to squamous cell carcinoma (SCC) comparing patients undergoing traditional symptomatic treatments with those patients that were treated by CO2 laser from 2004 - 2011. Outcome measures were rated by incisional biopsy (histology Report).

ELIGIBILITY:
Inclusion Criteria:

* Oral lichen planus
* Histological confirmation of diagnosis
* Patient willing for treatment

Exclusion Criteria:

* Patient just does not want to participate as control/study group

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 2004-01; Primary Completion 2011-11 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
stable disease of OLP (clinical observation) | 1 year

SECONDARY OUTCOMES:
Development of oral cancer (histological report after incisional biopsy) | 3 years

OTHER OUTCOMES:
Development of reccurrence of OLP (clinical observation) | 3 years